CLINICAL TRIAL: NCT06186401
Title: Phase 1 Study of Autologous Anti-EGFRvIII synNotch Receptor Induced Anti-EphA2/IL-13R alpha2 CAR (E-SYNC) T Cells in Adult Participants With EGFRvIII+ Glioblastoma
Brief Title: Anti-EGFRvIII synNotch Receptor Induced Anti-EphA2/IL-13Ralpha2 CAR (E-SYNC) T Cells
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hideho Okada, MD, PhD (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Hideho Okada, MD, PhD, Co-Principal Investigator, IND Holder, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23704; 5U19CA264338-03 (NIH)
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: EGFR Gene Mutation; Glioblastoma; MGMT-Unmethylated Glioblastoma; Recurrent Glioblastoma
Keywords: Immunotherapy; CAR T Therapy
MeSH Terms: conditions — Glioblastoma | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Starting Dose Level 1 (5 x 10^7 CAR+ cells) (DL1) (Experimental): Participants with newly diagnosed EGFRvIII+ GBM with unmethylated MGMT promotor status will undergo leukapheresis for manufacturing of E-SYNC T cells at least 2 weeks after completion of non-interventional, standard of care radiation therapy. Participants receive cyclophosphamide IV and fludarabine IV on days -5, -4, and -3 and then receive E-SYNC T cells IV on day 0. Participants will receive a single infusion of drug product (DP) (5 x 10^7 CAR+ T cells) and be monitored for safety, presence of and possible synNotch > CAR-T priming of the DP in the peripheral blood.
  Interventions: Biological: E-SYNC T Cells; Drug: Cyclophosphamide (non-investigational); Drug: Fludarabine (non-investigational); Procedure: Leukapheresis
- Cohort 1: Dose-escalation Level 2 (1.5 x 10^8 CAR+ cells) (DL2) (Experimental): If there are no dose-limiting toxicities in the starting dose cohort, participants with newly diagnosed EGFRvIII+ GBM with unmethylated MGMT promotor status will undergo leukapheresis for manufacturing of E-SYNC T cells at least 2 weeks after completion of tnon-interventional, standard of care radiation therapy. Participants receive cyclophosphamide IV and fludarabine IV on days -5, -4, and -3 and then receive E-SYNC T cells IV on day 0. Participants will receive a single infusion of drug product (DP) (1.5 x 10^8 CAR+ T cells) and be monitored for safety, presence of and possible synNotch > CAR-T priming of the DP in the peripheral blood.
  Interventions: Biological: E-SYNC T Cells; Drug: Cyclophosphamide (non-investigational); Drug: Fludarabine (non-investigational); Procedure: Leukapheresis
- Cohort 2: Tissue analysis cohort (Experimental): Participants with EGFRvIII+ glioblastoma recurrence after initial non-investigational, chemoradiation who need surgery will have the EGFRvIII H-scored based on digital image analysis of EGFRvIII immunohistochemistry (IHC) slides, with the score denoting both extent of and intensity of positive staining. Participants with an H-score of >=250 will undergo leukapheresis for manufacturing of E-SYNC T cells at the maximum tolerated dose, or recommended dose based on results from cohort 1 more than 2 weeks after completion of their non-investigational, standard of care radiation therapy. Participants will receive a single infusion of drug product (DP) on day 0 and will be admitted to the hospital for surgical resection (non-investigational) between days 14 and 28, and monitored for safety, presence of and possible synNotch > CAR-T priming of the DP in the peripheral blood, and anti-tumor response of E-SYNC T cells.
  Interventions: Biological: E-SYNC T Cells; Drug: Cyclophosphamide (non-investigational); Drug: Fludarabine (non-investigational); Procedure: Leukapheresis; Procedure: Surgical resection

INTERVENTIONS:
Biological: E-SYNC T Cells — Given IV
  Other Names: Anti-EGFRvIII synNotch Receptor Induced Anti-EphA2/IL-13R alpha2 CAR T Cells; Autologous Anti-EGFRvIII synNotch Receptor Induced Anti-EphA2/IL-13R alpha2 CAR T Cells; Autologous Anti-EGFRvIII synNotch Receptor Induced Anti-EphA2/IL-13Ra2 CAR T Cells
Drug: Cyclophosphamide (non-investigational) — Given IV
  Other Names: Cytoxan; Cytoxan Lyophilized; Neosar
Drug: Fludarabine (non-investigational) — Given IV
  Other Names: Fludara; Oforta
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Therapeutic Leukopheresis
Procedure: Surgical resection — Undergo surgical resection of tumor tissue
  Other Names: Resection
  Arms: Cohort 2: Tissue analysis cohort

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of E-SYNC chimeric antigen receptor (CAR) T cells after lymphodepleting chemotherapy in treating patients with EGFRvIII positive (+) glioblastoma. Chimeric antigen receptor (CAR) T-cell therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so the CAR T cells will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor. Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers. Lymphodepleting chemotherapy with cyclophosphamide and fludarabine before treatment with CAR T cells may make the CAR T cells more effective.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of IV infused E-SYNC T cells for the treatment of EGFRvIII positive (EGFRvIII+) glioblastoma (GBM) (both cohorts).

SECONDARY OBJECTIVES:

I. To evaluate the feasibility of production and administration of E-SYNC T cells for the treatment of GBM (both cohorts).

II. To determine the local priming of E-SYNC T cells by prospective evaluation of GBM tissue and peripheral blood (cohort 2 only).

EXPLORATORY OBJECTIVES:

I. To determine antitumor responses and survival after infusion of E-SYNC T cells.

II. To evaluate development of immune responses against E-SYNC T cells favoring rejection.

III. To characterize the intratumoral immune landscape.

OUTLINE: This is a dose-escalation study utilizing E-SYNC T cells.

COHORT 1 (Dose Escalation): An estimated 6 to 15 participants with newly diagnosed EGFRvIII+ glioblastoma with O6-methylguanine-DNA methyl-transferase (MGMT) unmethylated status who have completed initial radiation therapy will be assigned to cohort 1. Participants undergo leukapheresis for the creation of E-SYNC T cells at least 2 weeks after completion of their non-investigational, standard of care radiation therapy.

COHORT 2 (Tissue Cohort): An estimated 5-8 participants with EGFRvIII+ glioblastoma recurrence after initial chemoradiation who need surgery will be assigned to cohort 2. Participants undergo leukapheresis for the creation of E-SYNC T cells more than 2 weeks after completion of their non-interventional, standard of care radiation therapy. Participants also undergo standard of care (SOC) surgical resection.

After completion of study treatment, participants are followed up on days 1, 3, 7, 10, 14, 21, and 28, then every 4 weeks in weeks 8-24, every 8 weeks in weeks 32-48, every 12 weeks in weeks 60-96, every 3 months in months 24-36, and then annually in years 3-15.

NOTE: The product formulation has been adjusted as of Protocol Version 2.1. Due to this formulation change, the first 3 participants enrolled at DL 1 prior to the adjustment will not be counted towards dose escalation analysis. These participants will continue for safety evaluation. Starting with the 4th participant, new enrollees will receive the updated formulation and continue to enroll at DL 1 to ensure consistency in dosing escalation decisions. The 4th participant will therefore serve as the 1st participant in updated DL1 cohort. Hence, enrollment will be paused after 4th participant is treated in updated DL1 formulation and monitoring and subsequent infusions will proceed per the staggered schedule

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for Cohort 1:

  1. Age >= 18 years.
  2. Karnofsky performance status (KPS) score of >=70.
  3. All participants must have adequate organ function defined as:

     1. Peripheral absolute neutrophil count >=1000/mm^3.
     2. Platelet count >=100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
     3. Absolute lymphocyte count (ALC) >= 300/μL and/or Cluster of differentiation 3 (CD3) count of >=150/μL.
     4. Creatinine clearance or radioisotope glomerular filtration rate >= 50 mL/min/1.73m^2.
     5. Total Bilirubin <= 1.5 x ULN except for Gilbert's syndrome and
     6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 3x upper limit of normal (ULN).
     7. Left ventricular ejection fraction (LVEF) >= 40% by echocardiogram or multi-gated acquisition scanning (MUGA).
     8. Adequate pulmonary function, defined as no evidence of dyspnea at rest and pulse oximetry > 92% while breathing room air.
  4. Pathological criteria: EGFRvIII+ GBM from most recent surgery, confirmed by a Clinical Laboratory Improvement Amendments (CLIA)-certified lab using a next-generation sequencing panel.
  5. MGMT promoter must be unmethylated or with a methylation index < 3.
  6. Must have completed at least standard of care (SOC) external beam radiotherapy (EBRT) as initial therapy.
  7. Participants must be anticipated to be able to complete E-SYNC T cell infusion within 12 weeks after completion of EBRT.
  8. All participants must be off systemic steroids for 3 days or more prior to leukapheresis.
  9. Must be willing to provide voluntary informed consent for apheresis (and tissue screening if needed) and for study treatment.

NOTE: There are two sets of eligibility criteria for Cohort 2. Step 1 defines eligibility for tissue screening and apheresis, and Step 2 defines eligibility for study enrollment and E-SYNC T cell treatment.

* Inclusion Criteria for Cohort 2, Step 1:

  1. Age >=18 years.
  2. KPS score >=70.
  3. All participants must have adequate organ function defined as:

     1. Peripheral absolute neutrophil count >=1000/mm^3.
     2. Platelet count >=100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
     3. Absolute lymphocyte count (ALC) >= 300/μL and/or CD3 count of >=150/μL.
     4. Creatinine clearance or radioisotope glomerular filtration rate >= 50 mL/min/1.73m^2.
     5. Total Bilirubin <= 1.5 x ULN except for Gilbert's syndrome and
     6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 3x upper limit of normal (ULN).
     7. Left ventricular ejection fraction (LVEF) >= 40% by echocardiogram or multi-gated acquisition scanning (MUGA).
     8. Adequate pulmonary function, defined as no evidence of dyspnea at rest and pulse oximetry > 92% while breathing room air.
  4. Pathological criteria: EGFRvIII+ GBM from most recent surgery, as defined by an EGFRvIII + H-score of >=250 based on central review.
  5. All participants must be off systemic steroids for 3 days or more prior to leukapheresis.
  6. Must be willing to provide voluntary informed consent for apheresis (and tissue screening if needed).
* Inclusion Criteria for Cohort 2, Step 2. Note: Prior to Step 2, participants must have undergone leukapheresis in Step 1. In addition:

  1. KPS score >=70.
  2. Must have received at least SOC EBRT as initial therapy; any number of prior recurrences is allowed.
  3. Pathological criteria: EGFRvIII+ GBM from most recent surgery, as defined by an EGFRvIII + H-score of >=250 based on central review.
  4. Must have radiographic progression consistent with the Response assessment in neuro-oncology criteria (RANO) criteria for progressive disease (PD)
  5. Recurrence must be surgically amenable, with expectation for ability to resect at least 500mg of tumor tissue
  6. Participants with reproductive potential agree to use reliable and double barrier method of contraception during the study and for at least 6 months after the last study intervention, including refraining from donating sperm during this period.
  7. Females of childbearing potential must have a negative serum beta-Human Chorionic Gonadotropin (hCG) pregnancy test prior to receiving study interventions.
  8. All participants must have adequate organ function defined as:

     1. Peripheral absolute neutrophil count >=1000/mm^3.
     2. Platelet count >=100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
     3. Absolute lymphocyte count (ALC) >= 300/μL and/or CD3 count of >=150/μL.
     4. Creatinine clearance or radioisotope glomerular filtration rate >= 50 mL/min/1.73m^2.
     5. Total Bilirubin <= 1.5 x ULN except for Gilbert's syndrome and
     6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 3x upper limit of normal (ULN).
     7. Coagulation tests prothrombin time (PT) and partial thromboplastin time (PTT) have to be within normal limits, unless the participant has been therapeutically anticoagulated for previous venous thrombosis.
     8. Adequate pulmonary function, defined as no evidence of dyspnea at rest and pulse oximetry > 92% while breathing room air.
     9. Adequate cardiac function, confirmed within the last 12 months, defined as left ventricular ejection fraction (LVEF) >= 40% by echocardiogram or multi-gated acquisition scanning (MUGA).
  9. Must be willing to provide voluntary informed consent for apheresis (and tissue screening if needed).

Exclusion Criteria:

* Exclusion Criteria for Cohort 1

  1. Participant who has been treated with any investigational agents and chemotherapy targeting GBM <= 4 weeks prior to date of study registration. Exceptions to this include: must be >=23 days from last dose of temozolomide (TMZ) or radiotherapy, mush be >= 6 weeks from last dose of nitrosourea.
  2. Female participants of reproductive potential who are pregnant or lactating. Female study participants of reproductive potential must have a negative serum pregnancy test as part of eligibility confirmation.
  3. Known addiction to alcohol or illicit drugs.
  4. Prior treatment with any Epithelial Growth Factor Receptor (EGFR)-targeting therapy.
  5. Participants with leptomeningeal dissemination.
  6. Participants with a known disorder that affects their immune system, such as human immunodeficiency virus (HIV) or an autoimmune disorder requiring systemic cytotoxic or immunosuppressive therapy. Participants who are currently using non-systemic steroids (e.g., inhaled, intranasal, ocular, topical) are not excluded from the study.
  7. Participants with serologic status reflecting active hepatitis B or C infection. Participants that are positive for hepatitis B surface antigen (HBsAg+) will be excluded. Participants that are positive for hepatitis B core antibody or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. PCR positive participants will be excluded.
  8. Participants who have received prior solid organ or bone marrow transplantation.
  9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, second cancer currently receiving active treatment or anticipated to receive treatment within the next year, or psychiatric illness/social situations that would limit compliance with study requirements.
  10. Participants who are unable to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.
* Exclusion Criteria for Step 1 for Cohort 2

  1. Participant who has been treated with any investigational agents or chemotherapy targeting GBM <=4 weeks prior to date of study registration. Exceptions to this include: must be>= 23 days from last dose of TMZ or radiotherapy, must be>=6 weeks from last dose of nitrosourea.
  2. Female participants of reproductive potential who are pregnant or lactating. Female study participants of reproductive potential must have a negative serum pregnancy test as part of Step 1 eligibility confirmation.
  3. Uncontrolled active infection.
  4. Participants with a known disorder that affects their immune system, such as HIV or an autoimmune disorder requiring systemic cytotoxic or immunosuppressive therapy.

     Participants who are currently using non-systemic steroids (e.g., inhaled, intranasal, ocular, topical) are not excluded from the study.
  5. Participants with serologic status reflecting active hepatitis B or C infection. Participants that are positive for hepatitis B surface antigen (HBsAg+) will be excluded. Participants that are positive for hepatitis B core antibody or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. PCR positive participants will be excluded.
  6. Known addiction to alcohol or illicit drugs.
* Exclusion Criteria for Step 2 for Cohort 2

Prior to Step 2, participants must have undergone leukapheresis in Step 1. In addition:

1. Prior treatment with any EGFR-targeting therapy
2. Participant who has been treated with any investigational agents or chemotherapy targeting GBM <= 4 weeks prior to date of study registration. Exceptions to this include: must be >= 23 days from last dose of TMZ or radiotherapy, must be >= 6 weeks from last dose of nitrosourea.
3. Participants with imaging or clinical evidence of uncontrolled tumor mass effect; the assessment of mass effect will be made by the Investigators.
4. Participants with leptomeningeal dissemination.
5. Participants with a known disorder that affects their immune system, such as HIV or an autoimmune disorder requiring systemic cytotoxic or immunosuppressive therapy.

   Participants who are currently using inhaled, intranasal, ocular, topical, or other non-oral or non-IV steroids are not necessarily excluded from the study.
6. Participants with serologic status reflecting active hepatitis B or C infection. Participants that are positive for hepatitis B surface antigen (HBsAg+) will be excluded. Participants that are positive for hepatitis B core antibody or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. PCR positive participants will be excluded.
7. Participants who have received prior solid organ or bone marrow transplantation.
8. Female participants who are pregnant or breast-feeding.
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, second cancer currently receiving active treatment or anticipated to receive treatment within the next year, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Participants who are unable to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants reporting treatment-emergent adverse events | Up to 96 weeks
  Treatment-emergent adverse events will be graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0

SECONDARY OUTCOMES:
Percentage of participants who successfully receive E-SYNC T cells | Up to 96 weeks
  The percentage of participants for whom a sufficient quantity of drug product (E-SYNC T cells) could be manufactured from peripheral blood mononuclear cells (PBMC) obtained at apheresis and administered will be reported.
The percentage of primed E-SYNC T (Cohort 2 only) cells in TIL versus PBMC will be evaluated | Up to 96 weeks
  Success will be defined as at least 2 of the 5 (or 8) participants having an increase in primed E-SYNC T cells in tumor-infiltrating lymphocytes (TIL)vs PBMC of >= 15%

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Clarke, MD, MPH, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No